CLINICAL TRIAL: NCT06004219
Title: Peer Support in Patients With Diabetic Foot Ulceration
Brief Title: Peer Support for Patients With Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Casa Colina Hospital and Centers for Healthcare (Other)
Collaborators: University of Southern California (Other); Vascular Cures (Other); Department of Health and Human Services (U.S. Federal Agency); Rancho Los Amigos National Rehabilitation Center (Other)
Responsible Party: Principal Investigator, Emily Rosario, Executive Director, Casa Colina Hospital and Centers for Healthcare
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB:00002372
Record Dates: First submitted 2023-06-30; First posted 2023-08-22 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Foot Ulcer; Diabetic Wound; Diabetes Mellitus, Type 2; Diabetic Foot; Diabetes Complications; Peripheral Neuropathy
Keywords: numbness; tingling; muscle weakness; loss of balance; shooting pain
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2; Diabetes Complications; Peripheral Nervous System Diseases; Hypesthesia; Paresthesia; Muscle Weakness

STUDY DESIGN:
Intervention Model Description: We will assign 12 patients into peer support group (intervention) and 12 patients as control (usual care with no support group) group. Patients will be followed for 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Support Group (Experimental): Patients will be asked to complete a health-related quality of life (HRQOL) survey at enrollment, 3 months, and end of the study. Participants will complete the VascuQoL-6 and PROMIS in several domains of HRQOL (including global physical function, global mental function, fatigue, depression, sleep disturbance, pain behavior, and social satisfaction). Each participant will complete the PROMIS CAT tool on an iPad App and the data will be stored in the secure REDCap
  Interventions: Behavioral: Peer counseling group
- Usual Care Group (No Intervention): Subjects in this group will not participate in the peer group.

INTERVENTIONS:
Behavioral: Peer counseling group — A community advisory board (CAB) will be set up for need assessment and to design the peer support program. Virtual meetings will be held quarterly for year 1 and 2. The group will consist of (up to 12 members) and will include at least 2 patient partners (patients with a recently diagnosed ulcer), 2 peer pals (patients with a healed DFU), family members or caregivers (limited to only 1 person per family represented on the CAB), healthcare workers (podiatrist, nurse, or case manager), medical equipment company representatives, and others. We will ask them about potential barriers at the first meeting, have flexible meeting times, and intentionally limit the number of healthcare providers. At the last meeting, we will seek feedback and input from the CAB. In addition, this group will have the opportunity to participate in a focus group which will be moderated with a trained, bilingual assistant and will last 40-60 minutes.
  Arms: Peer Support Group

SUMMARY:
The objective of the study is to develop a peer support program that helps improve ulcer care in patients with a diabetic foot ulcer (DFU).Diabetes, peripheral arterial disease (PAD), foot ulceration, and subsequent amputation are unevenly patterned in terms of racial/ethnicity, socioeconomic status, health insurance, and geographic area. The project will identify opportunities to reduce health disparities among economically marginalized patients regarding DFU outcomes.

DETAILED DESCRIPTION:
Of the estimated 30 million people in the U.S. with diabetes, 34% will develop a DFU in their lifetime, and 50% of those with a DFU have concurrent PAD. Foot ulceration, which precedes 80% of amputations in diabetics, is associated with impaired physical function, reduced quality of life, and increased risk of death. Moreover, PAD, DFU, and subsequent major amputations are unevenly patterned in terms of racial/ethnic, SES, health insurance, and geographic status. More specifically, Black and Hispanic adults with an ischemic DFU have a higher prevalence of amputation than their White counterparts. The mechanisms of these observed disparities in amputation, beyond disease severity and comorbidities, are complex. However, evidence indicates that ulcer care (including wound care, diabetic shoe, offloading, and recognizing warning signs) is a significant challenge for low-income patients with an ischemic DFU. In addition, our team and other researchers have demonstrated how psychological, interpersonal, social, and healthcare system-level barriers limit appropriate ulcer and foot care. Furthermore, our qualitative data demonstrates a high rate of psychological and interpersonal factors to diabetic foot care that cannot be ignored. Clearly, there is a compelling need for innovative methods to improve DFU care that are based on health equity that led to diverse support. To address this gap, we propose a patient-centered and culturally tailored Peer-Pal Intervention (PPI) that helps promote ulcer care in patients with a DFU, while minimizing the burden placed on system resources.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* New ischemic DFU <6 months
* English or Spanish speaking
* Able to provide consent

Exclusion Criteria:

* incarceration or institutionalization
* unwillingness to participate in the PAI program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
VascuQoL-6 | Complete at enrollment visit
  A self-reported survey or questionnaire that facilitates health-related quality of life assessment in peripheral arterial disease. Each question is scored 1-4. The sum of each individual question is used to generate a "Total" Quality of Life Score. A higher value indicates better health status.
VascuQoL-6 | Complete at 3 month visit
  A self-reported survey or questionnaire that facilitates health-related quality of life assessment in peripheral arterial disease. Each question is scored 1-4. The sum of each individual question is used to generate a "Total" Quality of Life Score. A higher value indicates better health status.
VascuQoL-6 | Complete at 6 month visit, end of study
  A self-reported survey or questionnaire that facilitates health-related quality of life assessment in peripheral arterial disease. Each question is scored 1-4. The sum of each individual question is used to generate a "Total" Quality of Life Score. A higher value indicates better health status.
PROMIS (Patient Reported Outcomes Measurement Information System) | Complete at enrollment visit
  Set of person-centered measures which evaluates and monitors physical, mental and social health in adults. It will be administered using a computer adaptive test (CAT) where items are selected for administration from an item bank based upon the respondent's answers. Items are ordered by level of difficulty from low to high using the Item Response Theory. After a person provides a response, the estimated score is recalculated. The CAT continues to administer items until stopping rules are met. The stopping rules for adults are as follows: at least 4 items administered, 12-items are administered or the standard error is below a threshold (0.3 on the theta metric or 3.0 on the T-score metric).
PROMIS (Patient Reported Outcomes Measurement Information System) | Complete at 3 month visit
  Set of person-centered measures which evaluates and monitors physical, mental and social health in adults. It will be administered using a computer adaptive test (CAT) where items are selected for administration from an item bank based upon the respondent's answers. Items are ordered by level of difficulty from low to high using the Item Response Theory. After a person provides a response, the estimated score is recalculated. The CAT continues to administer items until stopping rules are met. The stopping rules for adults are as follows: at least 4 items administered, 12-items are administered or the standard error is below a threshold (0.3 on the theta metric or 3.0 on the T-score metric).
PROMIS (Patient Reported Outcomes Measurement Information System) | Complete at 6 month visit, end of study
  Set of person-centered measures which evaluates and monitors physical, mental and social health in adults. It will be administered using a computer adaptive test (CAT) where items are selected for administration from an item bank based upon the respondent's answers. Items are ordered by level of difficulty from low to high using the Item Response Theory. After a person provides a response, the estimated score is recalculated. The CAT continues to administer items until stopping rules are met. The stopping rules for adults are as follows: at least 4 items administered, 12-items are administered or the standard error is below a threshold (0.3 on the theta metric or 3.0 on the T-score metric).
Acceptability Questionnaire --Peer to Pal Intervention (PPI) | End of study, 6 month visit
  5-point scale: strongly agree, agree, neutral, disagree, and strongly disagree
Twenty Three Item Questionnaire (Heisler) | End of Study, 6 month visit
  The questionnaire is a follow-up patient assessment comprised of 23 questions derived and modified from (Heisler et al.) It is a series of open ended questions to evaluate the effectiveness and attitudes of peer support with participants who have diabetic foot ulcer.
Diabetes Distress Screening Scale (DDS17) | Complete at enrollment visit
  6-point scale: 1-not a problem, 2-slight problem, 3- moderate problem, 4-somewhat serious problem, 5-serious problem, 6-very serious problem. A mean item score of 3 or higher indicates a level of distress worthy of clinical attention.
Diabetes Distress Screening Scale (DDS17) | Complete at 3 month visit
  6-point scale: 1-not a problem, 2-slight problem, 3- moderate problem, 4-somewhat serious problem, 5-serious problem, 6-very serious problem. A mean item score of 3 or higher indicates a level of distress worthy of clinical attention.
Diabetes Distress Screening Scale (DDS17) | End of study, 6 month visit
  6-point scale: 1-not a problem, 2-slight problem, 3- moderate problem, 4-somewhat serious problem, 5-serious problem, 6-very serious problem. A mean item score of 3 or higher indicates a level of distress worthy of clinical attention.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rosario, PhD, Principal Investigator — Casa Colina Hospital and Centers for Healthcare
Locations (3):
- United States (3):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - University of Southern California, Los Angeles, California
  - Casa Colina Healthcare and Hospital, Pomona, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- [Result] Hoffstad O, Mitra N, Walsh J, Margolis DJ. Diabetes, lower-extremity amputation, and death. Diabetes Care. 2015 Oct;38(10):1852-7. doi: 10.2337/dc15-0536. Epub 2015 Jul 22. PMID 26203063
- [Result] Crocker RM, Palmer KNB, Marrero DG, Tan TW. Patient perspectives on the physical, psycho-social, and financial impacts of diabetic foot ulceration and amputation. J Diabetes Complications. 2021 Aug;35(8):107960. doi: 10.1016/j.jdiacomp.2021.107960. Epub 2021 May 23. PMID 34059410